CLINICAL TRIAL: NCT07373730
Title: Clinical and Radiographic Evaluation of the Efficacy of Injectable Platelet Rich Fibrin Mixed With Hyaluronic Acid in Treatment of Temporomandibular Joint Internal Derangement: A Randomized Controlled Trial
Brief Title: Evaluation of the Efficacy of Injectable Platelet-Rich Fibrin Mixed With Hyaluronic Acid in Treatment of Temporomandibular Joint Internal Derangement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/667
Record Dates: First submitted 2025-12-02; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-10

CONDITIONS: Temporomandibular Joint Disc Displacement
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator)
  Interventions: Drug: Hyalgan 20 mg in 2 ML Prefilled Syringe; Other: I-PRF
- control group (Active Comparator)
  Interventions: Drug: Hyalgan 20 mg in 2 ML Prefilled Syringe

INTERVENTIONS:
Drug: Hyalgan 20 mg in 2 ML Prefilled Syringe — For the control group: 1mm of the drug was injected into the joint. For the study group: 0.5mm of the drug was injected into the joint.
Other: I-PRF — Only given for the study group: 0.5mm of I-PRF was injected into the joint.
  Arms: study group

SUMMARY:
we inject I-PRF and Hyaluronic Acid inside the human TMJ with internal derangement after arthrocentesis, and follow-up is made to evaluate the effect of this treatment.

DETAILED DESCRIPTION:
This study was made to evaluate the efficacy of injectable Platelet Rich Fibrin (I-PRF) with Hyaluronic Acid (HA) injection after arthrocentesis in treatment of Temporomandibular joint Internal Derangement.

The study was conducted on 30 patients whose ages ranged from 18 to 40 years, presented with impaired jaw function, limited mouth opening, Pain during joint movement and clicking. TMJ internal derangement was verified by preoperative MRI.

Patients with MPDS only, systemic debilitating disease, previous surgery in the TMJ, previous arthrocentesis, previous trauma to the joint were excluded from the study.

Control group: 15 cases were treated by arthrocentesis then injection of 1ml of Hyaluronic acid (HA).

Study group: 15 cases were treated by arthrocentesis then injection of 0.5ml of Hyaluronic acid (HA) and 0.5ml of injectable platelet rich fibrin (I-PRF).

Clinical assessment of pain by VAS, clicking as present or not, maximum mouth opening in millimeters, right and left lateral movements and protrusive movements was done preoperatively and postoperatively at 1,3,6 months.

MRI assessment was done preoperatively and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged from 18 to 40 years old.
2. patients diagnosed with internal derangement of TMJ, suffering from limited mandibular movements, joint pain and clicking.
3. Patients who are free from any systemic disease (ASA I).

Exclusion Criteria:

1. Patients who have myofascial pain dysfunction syndrome only.
2. Patients who have previous surgery in TMJ.
3. Patients who have previous arthrocentesis within 1 year.
4. Patients with prosthetic joint replacement.
5. Patients allergic to any components of the injecting solution.
6. Patients who received previous trauma to the joint.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Maximum mouth opening | immediate preoperative then 1, 3 and 6 months postoperatively
  was measured in millimeters using a ruler or digital caliper. It is the vertical distance between the incisal edges of upper and lower central incisors at maximum opening while the patients were instructed to set in an upright position in a dental chair.
Lateral to Right movement | immediate preoperative then 1, 3 and 6 months postoperatively
  was measured in millimeters using a ruler or digital caliper. It is the horizontal distance between the maxillary and the mandibular midlines with the teeth slightly separated and the mandible moved towards the right side.
Lateral to Left movement | immediate preoperative then 1, 3 and 6 months postoperatively
  was measured in millimeters using a ruler or digital caliper. It is the horizontal distance between the maxillary and the mandibular midline with the teeth slightly separated and the mandible moved towards the left side.
Protrusive movement | immediate preoperative then 1, 3 and 6 months postoperatively
  was measured in millimeters using a ruler or digital caliper. It is the distance from midpoint of incisal edge of maxillary incisors to midpoint of incisal edge of the mandibular incisors during mandibular protrusion.
Joint Clicking | immediate preoperative then 1, 3 and 6 months postoperatively
  was measured in terms as present or absent by hearing and palpation over each joint during opening and closing jaw movements.
Joint Pain | immediate preoperative then 1, 3 and 6 months postoperatively
  was measured in a score from 0 to 10 using the visual analogue scale [VAS] over the TMJ area. [ 0 is given when there is no pain, 1-3 mild pain, 4-6 moderate pain, 7-9 severe pain, 10 the worst pain].

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Suez Canal University, Ismailia, Egypt